CLINICAL TRIAL: NCT01586871
Title: Carotid Structure and Function in MPS Syndromes: A Multicenter Study of the Lysosomal Disease Network
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); National Center for Advancing Translational Sciences (NCATS) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1202M09721; U54NS065768 (NIH)
Record Dates: First submitted 2012-04-25; First posted 2012-04-27 (Estimated); Results first posted 2021-02-03 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Mucopolysaccharidoses
Keywords: MPS I; MPS II; MPS IIIA; MPS VI
MeSH Terms: conditions — Mucopolysaccharidoses; Sudden Infant Death; Mucopolysaccharidosis III; Mucopolysaccharidosis VI

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Mucopolysaccharidosis (MPS) syndromes are disorders characterized by enzyme deficiencies, and they have been linked to heart health complications. However, there are currently no proven markers of heart and artery health for this population. The main purpose of this observational study is to evaluate the ease and convenience of a non-invasive measurement of artery function in MPS I, MPS II and MPS VI patients compared to healthy control subjects. An observational study is a research design meaning that there is no treatment in this study.

The research questions are:

1. Is the artery health of MPS I, II and VI patients different than healthy controls?
2. Is the artery health of MPS VI patients different than MPS I and II patients?

It is hypothesized that MPS patients will have poorer outcomes of artery health compared to healthy controls.

DETAILED DESCRIPTION:
Mucopolysaccharidosis (MPS) syndromes are disorders characterized by enzyme deficiencies. As a result of the enzyme deficiency, glycosaminoglycans that are normally recycled in a healthy individual cannot be degraded in the MPS patient. MPS syndromes have been linked to heart health complications. Complications related to coronary artery stenosis (narrowing) are recognized as potentially fatal sequelae of untreated and treated MPS. Presently, national guidelines are largely silent on coronary artery disease risk in this population. There are currently no validated markers of cardiovascular or coronary artery disease in the MPS population. The main purpose of this observational study is to evaluate the ease and convenience of a non-invasive measurement of artery function in MPS I, MPS II and MPS VI patients compared to healthy control subjects. Exploring the validity and usefulness of this non-invasive measurement is the first step towards developing validated markers of cardiovascular or coronary artery disease in the MPS population.

Specific Aim #1: Compare carotid artery intima-media thickness and carotid stiffness in individuals with MPS I, II, and VI (treated and non-treated) vs. healthy age-and gender-matched controls. It is hypothesized that MPS patients will have increased carotid artery thickness and reduced carotid compliance and distensibility compared to healthy controls.

Specific Aim #2: Compare carotid artery intima-media thickness and carotid stiffness in individuals with MPS VI vs. I and II and between MPS I patients clinically treated with HSCT vs. ERT. It is hypothesized that MPS VI will have decreased carotid thickness and increased carotid compliance and distensibility compared to MPS I and II and that MPS I patients treated with ERT will have increased carotid thickness and reduced carotid compliance and distensibility compared to MPS I patients treated with HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 3 and 18 years old
* Be diagnosed with MPS I, MPS II or MPS VI

Exclusion Criteria:

* None

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This is an observational study of 60 individuals with MPS I, II and VI between the ages of 3 and 18. Those participating in this study will be seen for a onetime, one-hour study visit. Participants will be enrolled at the University of Minnesota, Minneapolis, Minnesota and Children's Hospital of Orange County, Orange, California.
Sampling Method: Non-Probability Sample
Enrollment: 1147 (Actual)
Dates: Start 2012-03; Primary Completion 2016-08 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron S Kelly, Ph.D., Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - Children's Hospital of Orange County, Orange, California
  - University of Minnesota, Minneapolis, Minnesota

REFERENCES:
- See also: Rare Disease Clinical Research Network — https://rarediseasesnetwork.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a dual-center, cross-sectional assessment of carotid imaging data obtained from 33 patients with biochemically and/or molecularly confirmed MPS Types I, II, III and VI; 560 healthy pediatric control patients; and 554 adult control patients. The pediatric and adult controls were obtained from prior studies of insulin resistance and cardiovascular risk at the University of Minnesota. Clinical data from MPS patients were obtained from chart review.
Groups:
- Pediatric Control Patients: The pediatric control patients were obtained from prior studies of insulin resistance and cardiovascular risk at the University of Minnesota.
- Adult Controls: The adult controls were obtained from prior studies of insulin resistance and cardiovascular risk at the University of Minnesota.
- MPS Patients: Clinical data (demographic information, anthropometrics, ethnicity, confirmation of diagnosis, and treatment status) from MPS patients were obtained from chart review. For this project, data from MPS I, MPS II, MPS IIIa and MPS VI was available.
Period: Overall Study
Arm/Group | Pediatric Control Patients | Adult Controls | MPS Patients
Started | 560 | 554 | 33
Completed | 560 | 554 | 33
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pediatric Control: Healthy pediatric control subjects
- Adult Control: Healthy adult control subjects
- Mucopolysaccharidosis (MPS ) Subjects: Mucopolysaccharidosis subjects type I, II, IIIA and VI.
- Total: Total of all reporting groups
Arm/Group | Pediatric Control | Adult Control | Mucopolysaccharidosis (MPS ) Subjects | Total
Number analyzed (Participants) | 560 | 554 | 33 | 1147
Age, Continuous [Median (Standard Deviation); unit: years] | 13.14 (4.01) | 39.16 (2.24) | 12.47 (4.66) | 21.59 (3.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 259 | 285 | 10 | 554
  Male | 301 | 269 | 23 | 593
Height [Median (Standard Deviation); unit: centimeters] — measured in centimeters
  centimeters | 155 (18.3) | 171 (12.8) | 132 (16.59) | 152.66 (15.89)
Weight [Median (Standard Deviation); unit: kilograms] — measured in kilograms
  kilograms | 53.8 (23.54) | 86.39 (23.33) | 36.66 (16.74) | 58.95 (21.20)
Body Mass Index [Median (Standard Deviation); unit: Kg/m^2] | 21.44 (5.84) | 29.46 (7.47) | 20.03 (4.50) | 23.64 (5.93)
Systolic blood pressure [Median (Standard Deviation); unit: mm Hg] | 106 (10.42) | 125 (15.59) | 106 (10.98) | 112.33 (12.33)
Diastolic blood pressure [Median (Standard Deviation); unit: mm Hg] | 58 (7.78) | 71.97 (10.39) | 55 (13.73) | 61.65 (10.63)

OUTCOME MEASURES:

1. Primary Outcome: Carotid Intima-media Thickness, Measured in Millimeters
Description: The carotid intima-media thickness test (CIMT) is a measure used to diagnose the extent of carotid atherosclerotic vascular disease. The test measures the thickness of the inner two layers of the carotid artery-the intima and media-and alerts physicians to any thickening when patients are still asymptomatic. CIMT was measured from the far wall of the left common carotid.
Time Frame: Baseline
Measure: Median (Standard Deviation); unit: mm
Arm/Group | Pediatric Control | Adult Control | Mucopolysaccharidosis (MPS ) Subjects
Number analyzed (Participants) | 560 | 554 | 33
mm | 0.44 (0.04) | 0.52 (0.09) | 0.56 (0.05)

2. Secondary Outcome: Carotid Cross-sectional Distensibility
Description: Carotid distensibility is a measure of carotid artery elasticity that has been introduced as a risk factor for cardiovascular disease. It is defined by the percent change in carotid lumen area from diastole to systole, has the unit of % and is defined by the equation (sD^2 - dD^2/dD^2)*100 where sD is the maximum systolic carotid diameter, dD is the minimum diastolic carotid diameter. Increasing carotid distensibility reflects high carotid distensibility and low stiffness, and vice versa.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Pediatric Control | Adult Control | Mucopolysaccharidosis (MPS ) Subjects
Number analyzed (Participants) | 560 | 554 | 33
percentage of change | 32.03 (8.35) | 16.33 (4.73) | 28.36 (15.70)

3. Secondary Outcome: Carotid Cross-sectional Compliance
Description: This is defined by the relative change in carotid lumen area from diastole to systole for a given change in blood pressure, has the unit mm^2/mmHg and is defined by the equation ¶(sD^2-dD^2)/4*PP where PP is pulse pressure (or systolic blood pressure-diastolic blood pressure). Increasing carotid cross sectional compliance reflects high carotid distensibility and low stiffness, and vice versa.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mm^2*mm Hg-1
Arm/Group | Pediatric Control | Adult Control | Mucopolysaccharidosis (MPS ) Subjects
Number analyzed (Participants) | 560 | 554 | 33
mm^2*mm Hg-1 | 0.16 (0.05) | 0.11 (0.04) | 0.14 (0.08)

4. Secondary Outcome: Carotid Incremental Elastic Modulus
Description: A way of measuring the elasticity constant of the carotid vessel, has the unit mmHg and is defined by the equation 3(1+sD^2/dD^2)/cross sectional compliance value. In contrast to carotid cross sectional compliance and carotid cross sectional distensibility, increasing carotid incremental elastic modus reflects low carotid distensibility and high thickness.
Time Frame: Baseline
Measure: Median (Standard Deviation); unit: mm Hg
Arm/Group | Pediatric Control | Adult Control | Mucopolysaccharidosis (MPS ) Subjects
Number analyzed (Participants) | 560 | 554 | 33
mm Hg | 951 (379.84) | 1859 (755.3) | 1341 (817.06)

ADVERSE EVENTS:
Time Frame: This is a chart review study that collected data at only one timepoint.
Description: There were no adverse events to be reported as this is a chart review study.
Groups:
- MPS Patients: Individuals with MPS disease (17 MPS I, 9 MPS II, 4 MPS IIIA , 3 MPS VI)
- Pediatric Controls: Healthy pediatric control subjects
- Adult Controls: Healthy adult control subjects
Arm/Group | MPS Patients | Pediatric Controls | Adult Controls
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/560 | 0/554
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/560 | 0/554
Other Adverse Events (participants affected / at risk) | 0/33 | 0/560 | 0/554

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No